CLINICAL TRIAL: NCT03623295
Title: The Dynamic Interplay Between Bleeding Phenotype and Baseline Factor Level in Moderate and Mild Hemophilia A and B
Acronym: DYNAMO
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Karin Fijnvandraat, Professor of Pediatric Hematology, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL61564.018.17
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2021-10

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Blood Specimen Collection; Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Biospecimens to be retained for future research:
  * Blood
  * Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort study population: For the main cohort study, we will include 230 patients with moderate or mild hemophilia A or B.
  Interventions: Other: Blood sample; Other: Questionnaire
- Sub study population: A subset of 50 patients of the cohort study population will be investigated in more detail by longitudinal data collection.
  Interventions: Other: Blood sample; Other: MRI-imaging; Other: Physical examination

INTERVENTIONS:
Other: Blood sample — Blood withdrawal.
Other: Questionnaire — Online questionnaire about the bleeds that patients experienced in the past.
  Groups: Cohort study population
Other: MRI-imaging — MRI imaging of joints.
  Groups: Sub study population
Other: Physical examination — Physical examination of joint status.
  Groups: Sub study population

SUMMARY:
There are large inter-individual differences in the bleeding pattern of patients with moderate or mild hemophilia. The major determinant of bleeding phenotype is the level of coagulant factor VIII or IX. In hemophilia A, studies addressing the association between factor VIII level and the clinical bleeding pattern yield conflicting results. In hemophilia B such studies have not yet been performed.

The primary aim of this project is to analyze the association between factor VIII and factor IX levels and the bleeding phenotype. The secondary aim is to analyze potential differences in phenotype between hemophilia A and B.

The project is a multicentre observational cohort study. We will include 230 patients with moderate or mild hemophilia A or B (FVIII/FIX 0.02-0.35 IU/mL) who are 12 to 55 years old. The main cohort study consists of clinical data collection, one blood sample and an online questionnaire for patients. Data will be collected on the nature and duration of all bleeding episodes, disease and treatment characteristics, physical activity level and musculoskeletal status. One blood withdrawal will be performed for centralized laboratory assays for FVIII or FIX levels (both one-stage and chromogenic assays) and genetic analysis for the most prevalent prothrombotic mutations. The online questionnaire for patients focuses on bleeds experienced in the past.

A subset of 50 patients aged 24 years or older with mild and moderate hemophilia A will be investigated in more detail by longitudinal data collection including analysis of physical joint status, MRI imaging of joints and biomarkers for joint damage. This longitudinal observation will consist of two time points that lie two years apart, allowing us to identify any changes that occur over the observed time period with respect to joint status.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or mild hemophilia A (FVIII:C 0.02-0.35 IU/mL) or hemophilia B (FIX:C 0.02-0.35 IU/mL)
* Age from 12 up to and including 55 years

Exclusion Criteria:

* Other clotting disorder
* Participation in another trial with an investigational product
* Comorbidity affecting the musculoskeletal status
* Clinically relevant inhibitor status at present or in the past
* Hemophilia B Leyden
* Use of anticoagulants

Ages: 12 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients will be recruited from Hemophilia Treatment Centers participating in the INSIGHT consortium, a well-established and productive group of investigators from European countries, Canada and Australia.
Sampling Method: Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Bleeding phenotype | Retrospective 10 years
  Annual bleeding rate, annual major bleeding rate, annual spontaneous joint bleeding rate, annual joint bleeding rate

CONTACTS AND LOCATIONS:
Overall Officials: Karin Fijnvandraat, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (17):
- Royal Adelaide Hospital, Adelaide, Australia
- Medical University of Vienna, Vienna, Austria
- Multicentre: Leuven, Brussels, Multiple Locations, Belgium
- Multicentre: Vancouver, Toronto, Hamilton, Multiple Locations, Canada
- Helsinki University Central Hospital, Helsinki, Finland
- Multicentre: Bonn, Berlin, Frankfurt, München, Hamburg, Multiple Locations, Germany
- Multicentre: Florence, Rome, Parma, Milan, Turin, Multiple Locations, Italy
- Netherlands (8):
  - Academic Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - Utrecht University Medical Center, Utrecht
  - Máxima Medical Center, Veldhoven
- Multicentre: Valencia, Madrid, Barcelona, Multiple Locations, Spain
- Multicentre: Manchester, London, Liverpool, Glasgow, Cardiff, Sheffield, Multiple Locations, United Kingdom

IPD SHARING:
Plan to Share IPD: No